CLINICAL TRIAL: NCT02569567
Title: Applicability, Reliability and Accuracy for Staging Hepatic Fibrosis: Comparison of Smart-Shear Wave Elastography and Transient Elastography
Brief Title: Comparison of Smart-Shear Wave Elastography and Transient Elastography
Acronym: SMART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Assistant Professor, Asan Medical Center
Other Study IDs: SMART15; 2015-0782 (Other: Asan Medical Center Institution Review Board(IRB))
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-10

CONDITIONS: Fibrosis, Liver
Keywords: Smart-Shear Wave(SSW); Transient Elastography(TE); Liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- US elastography: Participants who have the plan of liver transplantation or liver biopsy within 4 weeks will be screened from the outpatient clinic.
  Two types of ultrasonographic elastography(US elastography) techniques including Smart-Shear Wave(SSW) imaging and transient elastography(TE) will be performed as a diagnostic method for hepatic fibrosis.
  Interventions: Procedure: Smart-Shear Wave(SSW) imaging; Procedure: Transient elastography(TE)

INTERVENTIONS:
Procedure: Smart-Shear Wave(SSW) imaging — 1. All Smart-Shear Wave(SSW) imaging examinations will be performed by one operator.
  2. The right lobe of the liver is examined through the intercostal view with the patient lying in a supine or semi-decubitus position with the right arm in maximal abduction.
  3. Once the optimal sizes of the regions of interest is chosen, they are fixed for subsequent measurement in each subject. Special attention is paid to avoid any focal lesion, vessels, biliary tracts, or artifacts from nearby lung gas or cardiac movement.
  Other Names: S-Shearwave
Procedure: Transient elastography(TE) — 1. Using the M probe in patients with BMI <30 kg/m2.
  2. Liver measurement is taken at either the seventh or eighth intercostal space of each subject over the right lobe of the liver. The measuring depth ranges from 2.5 to 6.5 cm below the skin surface.
  3. Examinations are performed by a sonographer blinded to S-shear wave elastography, and biological results.
  Other Names: FibroScan®

SUMMARY:
The aim of this prospective study was to evaluate the applicability and diagnostic performances of Smart-Shear wave(SSW) imaging, in comparison with Transient elastography(TE) for the staging of liver fibrosis using pathologic results as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with liver disease: plan to undergo liver surgery
2. Potential liver donors
3. Smart-Shear wave & transient elastography were performed within one month from liver surgery
4. Aged between 20 to 80 years
5. Compliance with scheduled visits, evaluation plans and other study procedures

Exclusion Criteria:

1. Previous history of hepatic surgery
2. Previous history of transarterial chemoembolization
3. Huge or infiltrative tumor in the right lobe of the liver
4. Bile duct dilatation in the right lobe of the liver
5. Older than 80 years
6. The opinion of the investigator would make the patient unsuitable for enrollment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 105 participants will be enrolled. Participants are patients with liver disease who are planning to undergo liver surgery, and potential liver donors for living related liver transplantation.
  Study population size was calculated by considering a power of 80%(1-sided alpha of 25%), and an expected dropout rate of 10%.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of Smart-Shear Wave(SSW) imaging compared to Transient elastography(TE) in diagnosis for hepatic fibrosis. | 1 year
  Applicability rate between Smart-Shear Wave(SSW) and Transient elastography(TE) will be compared to prove non-inferiority.
  Applicability rate = {[Total cases- (failure cases + non-reliable measurement cases)]/total case} * 100 (%)

SECONDARY OUTCOMES:
Evaluation of diagnostic accuracy to predict the degree of hepatic fibrosis. | 1 year
  Areas under the receiver operating curve (AUROCs) of the two techniques will be compared to estimate the probability of correctly predicting the degree of hepatic fibrosis.
  Substantial discordance between US elastography techniques and histologic staging will also be explored. It is defined as a difference in fibrosis stage by at least 2 points.
The correlation between two US elastography techniques | 1 year
  The correlation between the two US elastography techniques will be tested using the Spearman's correlation coefficient.
Reliability of Smart-Shear Wave(SSW) comparing diagnostic performance according to the reliable measurement index(RMI) results | 1 year
  Reliable measurement index (RMI) is an reliability index that computes the reliability of the calculated stiffness by analyzing the changes in shapes of propagated shear waves. The diagnostic performance of Smart-Shear wave will be assessed by comparing the RMI result.
Precision of Smart-Shear Wave(SSW) | 1 year
  Precision of Smart-Shear Wave(SSW) will be assessed using the composite factors, including intraclass correlation coefficients (ICCs), within subject SD(wSD), repeatability coefficient(RC), and within subject CV(wCV).

CONTACTS AND LOCATIONS:
Overall Officials: So Yeon Kim, Dr, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea